CLINICAL TRIAL: NCT04720014
Title: Enhancing Resilience in Senior Living Community Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Erickson Living Management, LLC (Unknown)
Responsible Party: Principal Investigator, Lara Traeger, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P002834
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Stress, Psychological; Coping Skills
Keywords: Resiliency; Flourishing; Coping Skills; Stress Reduction; Healthy Aging
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Single-arm, pre-test/post-test pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART-3RP Group Intervention (Experimental): Residents will participate in 9 structured weekly group sessions which incorporates stress management and relaxation training.
  Interventions: Behavioral: SMART-3RP Group Intervention

INTERVENTIONS:
Behavioral: SMART-3RP Group Intervention — Nine 1.5 hour group sessions focusing on developing:
  1. an understanding of stress physiology and the physiology of the relaxation response;
  2. a regular practice of eliciting the relaxation response; and
  3. cognitive behavioral and positive psychology/resilience skills.
  Participants receive a copy of the SMART-3RP session manual and audio recorded guided meditations for independent relaxation practice. Participants are encouraged to practice eliciting the relaxation response daily throughout the study, using the audio recordings or other mind body techniques. Participants will use a practice log to track their practice.

SUMMARY:
This single-arm pilot study tests the feasibility of integrating the Stress Management and Resiliency Training Relaxation Response Resiliency Program (SMART-3RP), a mind-body intervention, into senior living residential communities. The investigators hypothesize that the SMART-3RP intervention will be feasible for senior living community residents to attend.

ELIGIBILITY:
Inclusion Criteria:

* Resident of an Erickson Living senior living community
* Currently residing in an Erickson Living apartment home
* Sufficient English language skills to participate in study procedures

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unable or unwilling to participate in group sessions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
SMART-3RP group session attendance | Post-intervention (week 9)
  Percentage of participants who attend ≥6 of 9 sessions

SECONDARY OUTCOMES:
Resident satisfaction with participation in SMART-3RP intervention | Post-intervention (week 9)
  Proportion of participants who endorse satisfaction on individual survey items

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McEwen BS, Stellar E. Stress and the individual. Mechanisms leading to disease. Arch Intern Med. 1993 Sep 27;153(18):2093-101. PMID 8379800
- [Background] Population ageing and development: ten years after Madrid. Population Facts 2012/4. New York, NY: UN Dept of Economic and Social Affairs, Population Division; 2012. UN Dept of Economic and Social Affairs.
- [Background] Park ER, Traeger L, Vranceanu AM, Scult M, Lerner JA, Benson H, Denninger J, Fricchione GL. The development of a patient-centered program based on the relaxation response: the Relaxation Response Resiliency Program (3RP). Psychosomatics. 2013 Mar-Apr;54(2):165-74. doi: 10.1016/j.psym.2012.09.001. Epub 2013 Jan 22. PMID 23352048
- [Background] VanderWeele TJ. On the promotion of human flourishing. Proc Natl Acad Sci U S A. 2017 Aug 1;114(31):8148-8156. doi: 10.1073/pnas.1702996114. Epub 2017 Jul 13. PMID 28705870
- [Background] Park ER, Perez GK, Millstein RA, Luberto CM, Traeger L, Proszynski J, Chad-Friedman E, Kuhlthau KA. A Virtual Resiliency Intervention Promoting Resiliency for Parents of Children with Learning and Attentional Disabilities: A Randomized Pilot Trial. Matern Child Health J. 2020 Jan;24(1):39-53. doi: 10.1007/s10995-019-02815-3. PMID 31650412
- [Background] Gonzalez A, Shim M, Mahaffey B, Vranceanu AM, Reffi A, Park ER. The Relaxation Response Resiliency Program (3RP) in Patients with Headache and Musculoskeletal Pain: A Retrospective Analysis of Clinical Data. Pain Manag Nurs. 2019 Feb;20(1):70-74. doi: 10.1016/j.pmn.2018.04.003. Epub 2018 Dec 13. PMID 29773354
- [Background] Vranceanu AM, Riklin E, Merker VL, Macklin EA, Park ER, Plotkin SR. Mind-body therapy via videoconferencing in patients with neurofibromatosis: An RCT. Neurology. 2016 Aug 23;87(8):806-14. doi: 10.1212/WNL.0000000000003005. Epub 2016 Jul 22. PMID 27449066
- [Background] Stahl JE, Dossett ML, LaJoie AS, Denninger JW, Mehta DH, Goldman R, Fricchione GL, Benson H. Correction: Relaxation Response and Resiliency Training and Its Effect on Healthcare Resource Utilization. PLoS One. 2017 Feb 21;12(2):e0172874. doi: 10.1371/journal.pone.0172874. eCollection 2017. PMID 28222185
- [Background] Scult M, Haime V, Jacquart J, Takahashi J, Moscowitz B, Webster A, Denninger JW, Mehta DH. A healthy aging program for older adults: effects on self-efficacy and morale. Adv Mind Body Med. 2015 Winter;29(1):26-33. PMID 25607120
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Rounsaville BJ, Caroll KM, Onken LS. A stage model of behavioral therapies research: getting started and moving on from stage I. Clin Psychol Sci Pract. 2001;8:133-142.
- [Background] Shih WJ, Ohman-Strickland PA, Lin Y. Analysis of pilot and early phase studies with small sample sizes. Stat Med. 2004 Jun 30;23(12):1827-42. doi: 10.1002/sim.1807. PMID 15195318
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Derived] Traeger L, Styklunas GM, Park EY, Lee MT, Fricchione G, Park ER. Promoting Resilience and Flourishing Among Older Adult Residents in Community Living: A Feasibility Study. Gerontologist. 2022 Nov 30;62(10):1507-1518. doi: 10.1093/geront/gnac031. PMID 35235940